CLINICAL TRIAL: NCT06566365
Title: Effect of Hormonal Cahanges During Menstrual Cycle on Subcostal Transversus Abdominis
Brief Title: Effect of Hormonal Cahanges During Menstrual Cycle on Subcostal Transversus Abdominis Plane Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, MD, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADYU-ANS-NY-06
Record Dates: First submitted 2024-08-21; First posted 2024-08-22 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Menstrual Cycle; Subcostal Transversus Abdominis Plane Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group LB (Experimental): Patients that undergoing subcostal TAP block identified as being in the luteal phase by inquiring about the date of their last menstrual period.
  Interventions: Other: Subcostal Transversus Abdominis Plane Block
- Group FB (Experimental): Patients that undergoing subcostal TAP block identified as being in the follicular phase by inquiring about the date of their last menstrual period.
  Interventions: Other: Subcostal Transversus Abdominis Plane Block
- Group L (No Intervention): Patients identified as being in the luteal phase by inquiring about the date of their last menstrual period.
- Group F (No Intervention): Patients identified as being in the follicular phase by inquiring about the date of their last menstrual period.

INTERVENTIONS:
Other: Subcostal Transversus Abdominis Plane Block — After ensuring airway safety under general anesthesia, a bilateral Transversus Abdominis Plane Block using 20 cc of 0.25% bupivacaine with a subcostal approach under ultrasound guidance will be administered
  Arms: Group FB; Group LB

SUMMARY:
Fascial plane blocks are traditionally considered regional anesthesia techniques, where a mixture of local anesthetic (LA) is injected into a plane between two fascial layers, with the aim of spreading along this anatomical plane to block the nerves lying within or passing through it . Various pathophysiological processes that alter the structure and characteristics of fasciae can affect the spread of the local anesthetic and the success of the block. Diabetes, hormonal changes, and cannabinoid use are among these factors. This study aims to investigate the effects of hormonal changes during the menstrual cycle on subcostal TAP block.

DETAILED DESCRIPTION:
Female patients scheduled for laparoscopic cholecystectomy at Adıyaman University Training and Research Hospital, who have been informed about the study and have provided written consent to participate, will be included in the study. The patients who agree to participate will be divided into groups based on the phases of their menstrual cycles. After ensuring airway safety under general anesthesia, a bilateral TAP block using 20 cc of 0.25% bupivacaine with a subcostal approach under ultrasound guidance will be administered to both groups. The study aims to compare the hemodynamic values (arterial blood pressure, heart rate, peripheral oxygen saturation) during the perioperative period, the visual analog scale (VAS) scores postoperatively, and the Quality of Recovery-15 (QoR-15) scores at 24 hours postoperatively between the two groups. This will allow for the investigation of the effects of hormonal changes during the menstrual cycle on the efficacy and success of subcostal TAP blocks.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II, female, Laparoscopic cholecyctectomy, Subcostal TAP , 18-65 years old patient

Exclusion Criteria:

* ASA III-IV
* <18 , >65 years old patients
* menstrual disorders

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | postoperative 1st,2nd, 6.- 12.-24. hour
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Quality of Recovery - 15 | postoperative 24. hour
  The QoR-15 scale is a unidimensional measurement of quality of recovery measured in five domains: physical comfort, pain, physical independence, psychological support, and emotional state. The QoR-15 scale provides a score ranging from 0 to 150, with a high score indicating a good quality of recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No